CLINICAL TRIAL: NCT05006573
Title: A Multicentre, Randomised, Double-blind, Parallel-group, Placebo-controlled, 52 Week, Phase III Study With an Open-label Extension to Evaluate the Efficacy and Safety of Benralizumab in Patients With Non-Cystic Fibrosis Bronchiectasis (MAHALE)
Brief Title: Efficacy and Safety of Benralizumab in Patients With Non-cystic Fibrosis Bronchiectasis
Acronym: MAHALE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the decision to stop recruitment early, enrolment into the MAHALE trial was terminated in August 2022; 139 patients were screened and 100 randomised to IP.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D325BC00001; 2020-004068-24 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-08-16 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Benralizumab; Non-cystic Fibrosis Bronchiectasis; Eosinophlic Inflammation
MeSH Terms: interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab will be administered subcutaneously (SC) using an accessorized prefilled syringe (APFS)
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Matching placebo solution will be administered subcutaneously (SC) using an accessorized prefilled syringe (APFS)
  Interventions: Biological: Placebo to Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab active solution in a single accessorized prefilled syringe (APFS) will be administered subcutaneously (SC), 1 mL fill volume
  Arms: Benralizumab
Biological: Placebo to Benralizumab — Matching placebo solution in a single accessorized prefilled syringe (APFS) will be administered subcutaneously (SC), 1 mL fill volume
  Arms: Placebo

SUMMARY:
This is a multicentre, randomised, double-blind, parallel-group, placebo-controlled, phase III study originally designed to test the hypothesis that benralizumab will reduce exacerbation rates compared with placebo on top of standard-of-care therapy in adult patients with non-cystic fibrosis bronchiectasis with eosinophilic inflammation (NCFB+EI).

All patients who complete the double-blind treatment period (28 to 52 weeks depending on the timing of patient randomization and when the revised CSP version 3.0 becomes effective) on investigational product (IP) may be eligible to continue into an open-label extension (OLE) period during which all patients will receive benralizumab.

The revised OLE period is intended to allow patients approximately 32 weeks of treatment with open label benralizumab (24 weeks followed by a FU visit 8 weeks after the last dose of IP for a total of approximately 32 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age inclusive at the time of signing the ICF
* Must have NCFB diagnosed by a physician and confirmed by CT (measured at screening; if a new CT is not possible, a CT performed within 12 months of the screening visit is acceptable).
* Documented history of 2 or more bronchiectasis exacerbations within a year of the screening visit.
* If receiving prophylactic systemic or inhaled antibiotics to prevent bronchiectasis exacerbations, the dose/regimen must be stable for at least 3 months prior to the screening visit and remain stable throughout the DB period of the study. If prophylactic macrolides have been recently discontinued, patients must have been off treatment for at least 3 months prior to randomisation. In all other cases of prophylactic antibiotic use, ≥ 4 weeks wash out period should be in place after the last dose of antibiotic and prior to randomisation
* Must be on airway clearance therapy, physiotherapy, or mucus clearance therapy.The dose and regimen of these therapies and any drugs used to aid expectoration should be stable for at least 3 months prior to the screening visit and remain stable throughout the DB period of the study.
* If receiving inhaled corticosteroid or bronchodilator therapy, the dose and regimen should be stable with no alteration to dose or formulation for at least 3 months prior to the screening visit and this should remain stable throughout the DB period of the study.
* Women of childbearing potential (WOCBP) must have a negative serum and urine pregnancy test prior to randomization and agree to use a highly effective method of birth control from enrollment, throughout the study duration, and for 12 weeks after the last dose of IP.

Exclusion Criteria:

* Pulmonary disease other than bronchiectasis. Patients with a history of NTM disease may be enrolled if they have completed treatment prior to the Screening visit, if at least 3 months have elapsed since the last day of antibiotic treatment for NTM at the Screening visit, and if they have had a negative sputum culture prior to the screening visit.
* Another diagnosed or suspected pulmonary or systemic disease associated with elevated peripheral eosinophil counts
* Respiratory infection or bronchiectasis exacerbation during the screening period.
* Any other clinical condition that is not stable in the opinion of the Investigator and could:

  1. Affect the safety of the patient during the study.
  2. Influence the findings of the study or their interpretation.
  3. Impede the patient's ability to complete the entire duration of the study.
* Radiological findings suggestive of a respiratory disease other than bronchiectasis, suggestive of acute infection, or of solitary pulmonary nodules without appropriate follow up and demonstration of stability as per standard of care. Pulmonary nodules > 6 mm in size should have at least 2 years of follow up with no change on CT imaging.
* Current active liver disease
* Current malignancy, or history of malignancy, except for:

  1. Patients who have had basal cell carcinoma, localised squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided the patient is in remission and curative therapy was completed at least 12 months prior to Visit 1
  2. Patients who have had other malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years prior to Visit 1.
* History of known immunodeficiency disorder including a positive test for human immunodeficiency virus, HIV-1 or HIV-2.
* History of alcohol or drug abuse within the past year
* Current smokers with a tobacco history of ≥ 10 pack-years or ex-smoker with a tobacco history of ≥ 10 pack-years.
* Patients receiving long-term oxygen treatment
* Patients participating in, or scheduled for, an intensive (active) pulmonary rehabilitation programme. Patients who are in the maintenance phase of a rehabilitation programme are eligible.
* Use of non-invasive positive-pressure ventilation for conditions other than obstructive sleep apnoea
* Use of immunosuppressive medication within 3 months of the screening visit or expected need for chronic use (≥ 4 weeks) during study
* Receipt of any marketed or investigational biologic products (monoclonal or polyclonal antibody) within one year of the screening visit
* Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to randomisation
* Receipt of immunoglobulin and blood products within 30 days of the date of the screening visit
* Receipt of live attenuated vaccines within 30 days of the date of randomisation
* Concurrent enrolment in another clinical drug interventional trial
* History of anaphylaxis to any biologic therapy or vaccine
* Known history of allergy or reaction to any component of the IP formulation.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Judgement by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements
* Previous randomisation in the present study
* Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Chalmers, MD, Principal Investigator — University of Dundee, Nethergate, Dundee DD1 4HN, Scotland, UK
Locations (45):
- United States (4):
  - Research Site, Birmingham, Alabama
  - Research Site, Newport Beach, California
  - Research Site, Northridge, California
  - Research Site, El Paso, Texas
- Argentina (3):
  - Research Site, Florida
  - Research Site, San Fernando
  - Research Site, San Miguel de Tucumán
- Australia (2):
  - Research Site, Melbourne
  - Research Site, South Brisbane
- Canada (3):
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Windsor, Ontario
- China (3):
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Zhengzhou
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Hellerup
  - Research Site, Hvidovre
  - Research Site, Vejle
- Germany (4):
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Gauting
  - Research Site, München
- India (3):
  - Research Site, Coimbatore
  - Research Site, Hyderabad
  - Research Site, New Delhi
- Italy (4):
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Research Site, Quezon City, Philippines
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Penza
  - Research Site, Saratov
  - Research Site, Ulyanovsk
- South Korea (2):
  - Research Site, Jeonju
  - Research Site, Seoul
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Southampton, United Kingdom
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: MAHALE Poster Master US — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D325BC00001&attachmentIdentifier=61263d41-9ab6-4c9c-bea8-4c0d92e83002&fileName=941_MAHALE_Poster_V1.0_Master_US_enUS.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D325BC00001&attachmentIdentifier=d9d495e5-ee69-4191-918f-cbade8f6f117&fileName=d325bc00001-abbreviated-study-synopsis_Redacted_pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The plan was to randomize 420 eligible patients in a 1:1 ratio to receive either benralizumab or a matching placebo after screening. Patients were stratified at randomization by screening blood eosinophil category, country, and current chronic macrolide use. Due to the decision to stop recruitment early, 100 patients were randomized to receive benralizumab or placebo (20:80 in the low & high blood eosinophil strata). The revised DB treatment period was at least 28 weeks and up to 52 weeks.
Pre-assignment Details: All patients completed a screening period of 2 to 6 weeks during which inclusion/exclusion criteria was assessed, disease activity, lung function and patient reported outcomes (PROs) were recorded, medical history and clinical laboratory were taken.
Groups:
- Benralizumab 30 mg: Benralizumab 30 mg injection delivered subcutaneously every 4 weeks
- Placebo: Matching placebo injection delivered subcutaneously every 4 weeks
Period: Double-blind Treatment Period
Arm/Group | Benralizumab 30 mg | Placebo
Started | 54 | 45
Treated | 54 | 45
Completed | 42 | 42
Not Completed | 12 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Subject decision without consent withdrawn | 0 | 1
Period: Open-label Extension Period
Arm/Group | Benralizumab 30 mg | Placebo
Started (Not all double-blind participants enrolled in the Open-label extension period) | 38 | 40
Completed | 38 | 39
Not Completed | 0 | 1
Not completed — Subject decision without consent withdrawn | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received any Investigational Product were included in the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg | Placebo | Total
Number analyzed (Participants) | 54 | 45 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.14) | 59.2 (15.49) | 59.2 (14.18)
Age, Customized [Number; unit: participants]
  >= 18 to <= 65 years | 34 | 21 | 55
  > 65 years | 20 | 24 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 50 | 38 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 14 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 31 | 67
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bronchiectasis Exacerbations Rate in the Double-blind Period
Description: Annualized Non-Cystic Fibrosis Bronchiectasis (NCFB) exacerbations rate through end of double-blind treatment period.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: Full Analysis Set: All patients randomized and receiving at least one (1) dose of Investigational Product are included in the full analysis set, irrespective of their protocol adherence and continued participation in the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations per year
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
exacerbations per year | 1.44 [1.05 to 1.97] | 1.27 [0.89 to 1.80]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.5911, negative binomial model; marginal standardization method; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.71 to 1.82] — The rate ratio (Benralizumab/Placebo) and its 95% CI are estimated using a negative binomial model. The covariates include treatment arm, baseline blood eosinophil category, and number of exacerbations from previous year

2. Secondary Outcome: Time to First Exacerbation in the Double-blind Treatment Period
Description: Time to first NCFB exacerbation in the double-blind treatment period
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
days | 233 [118 to NA] — The upper limit of the median time to first exacerbation is not estimable due to insufficient number of participants with events. | 316 [141 to NA] — The upper limit of the median time to first exacerbation is not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6677, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.67 to 1.91] — The analysis is performed using cox proportional hazards model with covariates of treatment group, number of exacerbations in previous year and baseline eosinophil category

3. Secondary Outcome: Change From Baseline in QoL-B-RSS Over the Double-blind Period
Description: Change from baseline in Quality of Life-Bronchiectasis-Respiratory Symptoms Scale over the double-blind treatment period. QoL-B-RSS scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 6.6 (12.57) | 3.1 (11.65)
  Week 4 | 5.8 (12.53) | -1.5 (12.49)
  Week 6 | 6.8 (14.39) | 0.7 (10.94)
  Week 8 | 6.6 (14.17) | 2.1 (16.29)
  Week 10 | 5.3 (13.02) | -1.0 (14.46)
  Week 12 | 7.2 (11.47) | 0.9 (15.44)
  Week 14 | 8.0 (12.28) | 3.7 (14.63)
  Week 16 | 6.2 (14.51) | 1.3 (15.79)
  Week 18 | 8.6 (14.41) | 2.6 (18.60)
  Week 20 | 8.6 (15.41) | 1.4 (18.58)
  Week 22 | 8.4 (13.30) | 3.9 (20.33)
  Week 24 | 9.3 (17.31) | 4.4 (17.70)
  Week 26 | 7.4 (15.07) | 3.8 (18.40)
  Week 28 | 6.5 (15.92) | 2.7 (21.33)
  Week 30 | 7.5 (14.26) | 1.2 (17.32)
  Week 32 | 12.1 (14.37) | 2.4 (19.09)
  Week 34 | 7.6 (12.58) | 2.8 (18.90)
  Week 36 | 9.6 (17.44) | 3.6 (19.31)
  Week 38 | 8.1 (14.96) | 1.3 (17.68)
  Week 40 | 9.6 (17.32) | -1.1 (18.50)
  Week 42 | 7.1 (14.93) | 3.3 (16.25)
  Week 44 | 7.5 (15.00) | 0.8 (20.76)
  Week 46 | 8.6 (17.76) | 3.4 (18.89)
  Week 48 | 8.1 (16.75) | 3.2 (20.52)
  Week 50 | 9.8 (14.63) | 0.1 (15.42)
  Week 52 | 7.3 (17.91) | 0.2 (18.12)

4. Secondary Outcome: Change From Baseline in Pre-dose Pre-BD FEV1 Over the Double-blind Treatment Period
Description: Change from baseline in pre-dose pre-bronchodilator (BD) forced expiratory volume in one second (FEV1) over the double-blind treatment period
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
L
  Week 4 | 0.0139 (0.14327) | -0.0477 (0.10758)
  Week 8 | 0.0048 (0.15392) | -0.0465 (0.15263)
  Week 16 | -0.0191 (0.15964) | -0.0282 (0.11452)
  Week 24 | -0.0378 (0.17290) | -0.0595 (0.16409)
  Week 32 | -0.0248 (0.16782) | -0.0921 (0.17543)
  Week 40 | -0.0597 (0.18924) | -0.1037 (0.16808)
  Week 48 | -0.1236 (0.16353) | -0.0849 (0.13783)
  Week 52 | -0.1093 (0.13130) | -0.1186 (0.14969)

5. Secondary Outcome: Change From Baseline in LCQ Total Score Over the Double-blind Period
Description: Change from baseline in Leicester Cough Questionnaire (LCQ) total score over the double-blind treatment period. LCQ total scores range from 3 to 21. Higher scores indicate better quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 0.5 (2.22) | 0.5 (2.13)
  Week 4 | 0.7 (2.35) | 0.0 (2.15)
  Week 6 | 0.8 (2.76) | 0.6 (2.56)
  Week 8 | 0.8 (3.37) | 0.3 (2.85)
  Week 10 | 1.0 (2.77) | 0.1 (2.76)
  Week 12 | 1.0 (2.51) | 0.4 (3.03)
  Week 14 | 1.4 (2.78) | 0.8 (3.16)
  Week 16 | 0.9 (2.61) | 0.5 (3.10)
  Week 18 | 1.0 (3.42) | 1.1 (3.55)
  Week 20 | 1.4 (3.28) | 0.8 (3.39)
  Week 22 | 0.9 (3.32) | 0.8 (4.03)
  Week 24 | 1.0 (3.43) | 1.2 (3.48)
  Week 26 | 0.9 (3.58) | 1.0 (3.54)
  Week 28 | 0.5 (4.31) | 0.9 (4.08)
  Week 30 | 0.7 (3.33) | 0.8 (4.06)
  Week 32 | 1.8 (3.45) | 0.7 (4.14)
  Week 34 | 0.8 (2.43) | 0.8 (3.92)
  Week 36 | 1.2 (3.48) | 0.8 (3.95)
  Week 38 | 1.0 (3.61) | 0.6 (4.24)
  Week 40 | 1.2 (3.93) | 0.2 (3.86)
  Week 42 | 0.6 (3.42) | 0.3 (4.19)
  Week 44 | 0.5 (3.23) | 0.3 (4.02)
  Week 46 | 0.7 (3.68) | 0.6 (4.22)
  Week 48 | 0.3 (3.78) | 0.5 (4.20)
  Week 50 | 0.7 (3.29) | -0.2 (3.41)
  Week 52 | 0.2 (3.94) | -0.1 (2.86)

6. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Physical Functioning Scale
Description: change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Physical Functioning Scale. QoL-B Physical Functioning Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 0.5 (12.23) | -0.0 (16.50)
  Week 4 | 1.5 (17.68) | 0.8 (19.39)
  Week 6 | 4.1 (20.81) | 0.2 (17.97)
  Week 8 | 3.3 (15.07) | 0.3 (20.81)
  Week 10 | 1.5 (19.22) | 1.0 (22.06)
  Week 12 | 3.1 (19.54) | 0.5 (21.89)
  Week 14 | 4.4 (15.48) | 4.2 (22.15)
  Week 16 | 3.5 (18.06) | 3.3 (25.17)
  Week 18 | 4.8 (19.15) | 2.2 (23.01)
  Week 20 | 4.5 (18.45) | 4.7 (25.18)
  Week 22 | 3.1 (19.62) | 2.2 (22.96)
  Week 24 | 5.2 (18.21) | 4.7 (23.03)
  Week 26 | 3.6 (20.68) | 3.6 (24.40)
  Week 28 | 3.8 (24.77) | 4.8 (24.39)
  Week 30 | 2.5 (21.33) | 4.8 (25.50)
  Week 32 | 6.7 (18.80) | 5.9 (24.73)
  Week 34 | 2.7 (19.14) | 3.5 (24.90)
  Week 36 | 0.6 (22.76) | 4.7 (24.78)
  Week 38 | 1.9 (16.40) | 3.5 (23.5)
  Week 40 | 2.1 (23.55) | 4.1 (25.01)
  Week 42 | 1.3 (21.13) | 5.5 (28.92)
  Week 44 | 0.6 (23.62) | 4.2 (24.03)
  Week 46 | 2.0 (22.89) | 7.9 (23.42)
  Week 48 | 0.0 (27.89) | 7.6 (22.98)
  Week 50 | 5.3 (23.46) | 1.3 (21.08)
  Week 52 | 5.1 (23.90) | 2.1 (19.25)

7. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Role Functioning Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Role Functioning Scale. QoL-B Role Functioning Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 1.1 (13.64) | -1.2 (11.11)
  Week 4 | 2.8 (13.00) | -0.3 (14.53)
  Week 6 | 2.7 (14.80) | 2.5 (12.05)
  Week 8 | 0.5 (16.27) | 0.2 (15.02)
  Week 10 | 1.2 (14.09) | 2.7 (16.32)
  Week 12 | 1.7 (16.36) | 2.3 (16.96)
  Week 14 | 3.0 (16.10) | 2.1 (16.70)
  Week 16 | 0.1 (17.77) | -0.3 (16.60)
  Week 18 | 2.4 (16.93) | -0.0 (17.67)
  Week 20 | 0.9 (16.01) | 0.5 (18.25)
  Week 22 | 2.8 (21.11) | 4.0 (20.47)
  Week 24 | 1.9 (22.60) | 0.6 (19.67)
  Week 26 | -0.1 (21.44) | 1.2 (18.36)
  Week 28 | -1.9 (21.02) | 2.7 (17.79)
  Week 30 | 1.1 (20.83) | -0.3 (19.04)
  Week 32 | 4.4 (15.08) | 0.2 (18.17)
  Week 34 | 1.4 (18.01) | 1.7 (17.97)
  Week 36 | -0.6 (19.18) | 0.5 (16.69)
  Week 38 | 1.4 (18.15) | -2.2 (19.65)
  Week 40 | 1.7 (22.20) | 0.2 (21.80)
  Week 42 | -1.3 (21.48) | 1.8 (20.19)
  Week 44 | 0.6 (25.33) | -1.4 (17.46)
  Week 46 | 0.4 (23.89) | 4.0 (19.00)
  Week 48 | -1.2 (25.03) | 0.2 (18.16)
  Week 50 | 0.7 (21.26) | -1.9 (12.55)
  Week 52 | -0.8 (23.28) | 1.1 (17.81)

8. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Emotional Functioning Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Emotional Functioning Scale. QoL-B Emotional Functioning Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 0.2 (13.63) | 2.0 (17.43)
  Week 4 | -0.7 (14.07) | 1.4 (14.42)
  Week 6 | 3.5 (17.99) | 4.2 (14.98)
  Week 8 | -1.2 (16.84) | 1.4 (17.77)
  Week 10 | 0.2 (16.43) | -1.0 (16.58)
  Week 12 | 2.8 (17.30) | 1.6 (21.38)
  Week 14 | 4.7 (14.31) | 1.8 (20.79)
  Week 16 | 2.2 (16.56) | 1.2 (22.48)
  Week 18 | 3.2 (15.57) | 3.8 (21.68)
  Week 20 | 3.9 (15.82) | 1.4 (22.27)
  Week 22 | 2.8 (18.46) | 2.1 (23.09)
  Week 24 | 2.4 (17.80) | 2.9 (19.32)
  Week 26 | 3.0 (17.15) | 4.3 (22.00)
  Week 28 | 0.4 (25.82) | 1.6 (24.43)
  Week 30 | 2.7 (22.55) | 1.5 (23.79)
  Week 32 | 4.0 (15.82) | 3.0 (22.42)
  Week 34 | 1.4 (19.64) | 1.9 (23.23)
  Week 36 | 1.9 (17.89) | 4.5 (22.75)
  Week 38 | 2.6 (20.79) | 1.9 (22.64)
  Week 40 | 1.7 (23.35) | 2.3 (22.28)
  Week 42 | 1.1 (21.97) | 3.4 (22.67)
  Week 44 | 1.9 (25.89) | 1.8 (18.95)
  Week 46 | 3.9 (22.02) | 6.8 (22.77)
  Week 48 | 5.8 (22.10) | 5.4 (22.83)
  Week 50 | 5.5 (20.69) | 3.0 (18.14)
  Week 52 | 6.0 (26.30) | 0.9 (24.98)

9. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Social Functioning Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Social Functioning Scale. QoL-B Social Functioning Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 6.4 (17.60) | 4.5 (17.35)
  Week 4 | 4.4 (18.62) | 6.3 (22.69)
  Week 6 | 8.4 (21.60) | 5.8 (20.05)
  Week 8 | 9.7 (23.10) | 9.2 (20.53)
  Week 10 | 9.4 (19.64) | 6.0 (20.31)
  Week 12 | 10.6 (23.32) | 5.8 (21.42)
  Week 14 | 10.9 (23.03) | 7.7 (20.52)
  Week 16 | 9.1 (20.73) | 6.0 (23.53)
  Week 18 | 11.6 (21.61) | 10.3 (22.43)
  Week 20 | 11.8 (22.59) | 8.9 (21.43)
  Week 22 | 7.2 (20.42) | 9.5 (24.09)
  Week 24 | 10.1 (24.90) | 10.7 (24.14)
  Week 26 | 10.1 (22.86) | 9.9 (22.46)
  Week 28 | 8.8 (24.67) | 8.7 (24.83)
  Week 30 | 10.2 (26.57) | 7.7 (24.82)
  Week 32 | 12.8 (23.84) | 8.6 (24.48)
  Week 34 | 9.6 (27.93) | 9.3 (24.95)
  Week 36 | 12.0 (27.06) | 8.1 (25.53)
  Week 38 | 10.2 (27.83) | 6.5 (25.41)
  Week 40 | 13.9 (32.35) | 8.3 (27.77)
  Week 42 | 10.2 (29.40) | 8.6 (28.16)
  Week 44 | 9.9 (28.68) | 1.8 (24.50)
  Week 46 | 9.1 (27.40) | 6.6 (29.11)
  Week 48 | 12.1 (27.11) | 3.9 (30.74)
  Week 50 | 10.2 (23.60) | -1.7 (26.85)
  Week 52 | 11.6 (27.91) | 2.3 (25.29)

10. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Vitality Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Vitality Scale. QoL-B Vitality Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 3.0 (18.77) | -2.4 (13.54)
  Week 4 | 3.1 (17.82) | 0.3 (15.21)
  Week 6 | 4.0 (18.83) | -2.0 (13.88)
  Week 8 | 4.9 (17.84) | -1.1 (16.26)
  Week 10 | 6.4 (16.32) | -3.1 (18.83)
  Week 12 | 5.8 (18.48) | -3.9 (16.24)
  Week 14 | 8.8 (20.69) | -2.7 (18.22)
  Week 16 | 5.2 (19.66) | -0.5 (19.71)
  Week 18 | 5.0 (19.78) | -1.4 (18.69)
  Week 20 | 7.1 (19.99) | -1.3 (19.28)
  Week 22 | 5.7 (21.66) | -0.6 (21.04)
  Week 24 | 4.1 (20.87) | 1.0 (19.67)
  Week 26 | 6.2 (20.18) | -1.6 (20.66)
  Week 28 | 3.9 (21.75) | -2.1 (21.57)
  Week 30 | 4.4 (21.84) | -4.3 (22.74)
  Week 32 | 6.1 (19.97) | 0.0 (20.49)
  Week 34 | 1.1 (18.98) | -0.8 (20.96)
  Week 36 | 1.0 (18.59) | -2.7 (18.72)
  Week 38 | 4.1 (18.88) | -0.0 (19.52)
  Week 40 | 2.6 (23.01) | -2.7 (21.97)
  Week 42 | 3.0 (21.54) | -1.0 (24.37)
  Week 44 | 2.9 (21.11) | -3.4 (21.24)
  Week 46 | 5.2 (24.65) | 1.0 (20.10)
  Week 48 | 2.0 (23.48) | -1.3 (20.97)
  Week 50 | 7.7 (20.81) | 0.0 (18.14)
  Week 52 | 5.3 (18.74) | -5.3 (23.53)

11. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Health Perceptions Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Health Perceptions Scale. QoL-B Health Perceptions Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 1.3 (12.95) | 3.3 (14.12)
  Week 4 | 1.2 (14.87) | -0.2 (16.72)
  Week 6 | 3.5 (16.90) | 3.7 (16.06)
  Week 8 | 5.3 (17.23) | 4.3 (18.46)
  Week 10 | 5.6 (16.57) | 2.1 (18.47)
  Week 12 | 7.5 (16.69) | 3.3 (17.74)
  Week 14 | 7.4 (16.78) | 1.4 (18.99)
  Week 16 | 1.9 (16.25) | 2.4 (20.35)
  Week 18 | 5.8 (16.68) | 1.7 (20.69)
  Week 20 | 4.6 (18.21) | 3.9 (21.70)
  Week 22 | 5.0 (16.70) | 6.3 (21.99)
  Week 24 | 7.2 (17.18) | 5.0 (19.85)
  Week 26 | 2.8 (16.76) | 5.0 (20.26)
  Week 28 | 3.4 (18.81) | 2.4 (20.68)
  Week 30 | 4.5 (18.03) | 4.3 (21.87)
  Week 32 | 7.0 (16.37) | 2.4 (20.09)
  Week 34 | 4.2 (17.68) | 2.9 (22.29)
  Week 36 | 3.5 (17.84) | 2.0 (20.56)
  Week 38 | 4.2 (16.30) | 3.0 (22.90)
  Week 40 | 5.1 (16.95) | 1.4 (22.35)
  Week 42 | 4.7 (18.38) | 4.4 (23.77)
  Week 44 | 4.8 (21.03) | 1.5 (20.78)
  Week 46 | 6.6 (22.45) | 1.8 (19.07)
  Week 48 | 7.3 (21.32) | 3.9 (23.68)
  Week 50 | 6.9 (20.42) | 4.7 (18.65)
  Week 52 | 4.0 (21.53) | 0.4 (24.13)

12. Secondary Outcome: Change From Baseline in QoL-B Scales (Excluding QoL-B-RSS) Over the Double-blind Period: Treatment Burden Scale
Description: Change from baseline in Quality of Life-Bronchiectasis (QoL-B) scales (excluding QoL-B-RSS) over the double-blind treatment period: Treatment Burden Scale. QoL-B Treatment Burden Scale scores range from 0 to 100, with higher scores indicative of better health-related quality of life.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 2 | 3.6 (22.56) | -2.2 (16.75)
  Week 4 | 3.7 (18.62) | -2.1 (13.34)
  Week 6 | 6.0 (23.20) | -2.1 (15.72)
  Week 8 | 4.8 (18.35) | -1.9 (14.87)
  Week 10 | 4.0 (17.31) | 1.1 (17.83)
  Week 12 | 0.3 (17.27) | -0.4 (12.54)
  Week 14 | 0.6 (20.74) | -4.1 (14.73)
  Week 16 | 4.4 (20.10) | -1.1 (16.34)
  Week 18 | -1.9 (16.28) | -1.2 (14.92)
  Week 20 | 4.1 (16.01) | 0.3 (15.84)
  Week 22 | -1.3 (14.37) | -0.8 (16.82)
  Week 24 | -1.0 (18.58) | -1.1 (14.45)
  Week 26 | 1.9 (17.32) | 2.5 (15.37)
  Week 28 | -5.1 (24.00) | 1.4 (15.11)
  Week 30 | -2.0 (19.14) | -1.1 (18.39)
  Week 32 | -2.1 (16.32) | -0.8 (15.12)
  Week 34 | -0.4 (16.70) | -4.0 (17.95)
  Week 36 | -0.7 (16.68) | -1.5 (16.69)
  Week 38 | -4.2 (25.27) | -2.9 (21.04)
  Week 40 | -2.0 (24.76) | -0.4 (16.15)
  Week 42 | -1.5 (23.52) | 1.7 (18.78)
  Week 44 | 2.1 (17.22) | 1.4 (21.00)
  Week 46 | -0.0 (18.59) | 4.6 (14.62)
  Week 48 | -0.9 (17.25) | 3.6 (19.96)
  Week 50 | -2.0 (22.13) | -1.9 (18.77)
  Week 52 | -1.9 (25.64) | 1.7 (14.94)

13. Secondary Outcome: Change From Baseline in SGRQ Total Score Over the Double-blind Treatment Period
Description: Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score over the double-blind treatment period. SGRQ total scores range from 0 to 100. 100 represents the worst possible health status and 0 indicates the best possible health status.
Time Frame: through Double-blind period, at least 28 weeks and up to 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 54 | 45
score on a scale
  Week 4 | -4.7 (14.92) | 0.6 (14.89)
  Week 8 | -4.3 (15.99) | -2.4 (15.33)
  Week 16 | -4.4 (15.03) | -0.1 (16.06)
  Week 24 | -6.3 (16.21) | -3.9 (21.08)
  Week 32 | -5.8 (15.73) | -1.6 (21.46)
  Week 40 | -5.8 (17.63) | -1.6 (24.51)
  Week 48 | -4.9 (18.58) | -0.0 (22.45)
  Week 52 | -4.4 (20.37) | 4.8 (23.33)

ADVERSE EVENTS:
Time Frame: Double-Blind Treatment Period: From first dose of study drug until end of double-blind period, up to 52 weeks. Open-label Extension Period: From the end of the double-blind period (week 25 to 53) to the end of open-label extension period, up to 40 weeks.
Description: For analysis of Adverse Events, Safety Analysis Set is used. Safety Analysis Set: All participants who received at least one dose of study drug.
Groups:
- Benra 30 mg - DB: Benralizumab 30 mg injection delivered subcutaneously every 4 weeks, Double-blind period
- Placebo - DB: Matching placebo injection delivered subcutaneously every 4 weeks, Double-blind period
- Benra 30 mg - OLE: Benralizumab injections delivered subcutaneously every 4 weeks, Open-label extension period (Participants who took Double-blind benralizumab previously)
- Placebo Swithed to Benra 30 mg - OLE: Benralizumab injections delivered subcutaneously every 4 weeks, Open-label extension period (Participants who took Double-blind placebo previously)
Arm/Group | Benra 30 mg - DB | Placebo - DB | Benra 30 mg - OLE | Placebo Swithed to Benra 30 mg - OLE
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/45 | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 10/54 | 3/45 | 5/38 | 4/40
Other Adverse Events (participants affected / at risk) | 33/54 | 18/45 | 9/38 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg - DB (N=54) | Placebo - DB (N=45) | Benra 30 mg - OLE (N=38) | Placebo Swithed to Benra 30 mg - OLE (N=40)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (4) | 2 (2) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg - DB (N=54) | Placebo - DB (N=45) | Benra 30 mg - OLE (N=38) | Placebo Swithed to Benra 30 mg - OLE (N=40)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 5 (7) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 18 (18) | 10 (11) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (8) | 5 (5) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT05006573/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT05006573/SAP_001.pdf